CLINICAL TRIAL: NCT05623345
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase 2b/3 Study to Evaluate the Efficacy and Safety of Izokibep in Subjects With Active Psoriatic Arthritis
Brief Title: Psoriatic Arthritis Study of Izokibep
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Per our 13Aug24 press release, we announced discontinuation of internal development in this indication. This decision was not due to safety reasons.
Sponsor: ACELYRIN Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22104; 2022-501362-22 (Other: EU Trial Number)
Record Dates: First submitted 2022-11-13; First posted 2022-11-21 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-11

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis (PsA); psoriasis; inflammatory arthritis; enthesitis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Placebo from Day 1/Week 0 to Week 15, then izokibep from Week 16 to Week 51
  Interventions: Drug: Izokibep; Drug: Placebo to izokibep
- Group 2 (Experimental): Izokibep Dose 1 from Day 1/Week 0 to Week 51
  Interventions: Drug: Izokibep
- Group 3 (Experimental): Izokibep Dose 2 from Day 1/Week 0 to Week 51
  Interventions: Drug: Izokibep; Drug: Placebo to izokibep
- Group 4 (Experimental): Izokibep Dose 3 from Day 1/Week 0 to Week 51
  Interventions: Drug: Izokibep; Drug: Placebo to izokibep

INTERVENTIONS:
Drug: Izokibep — Biologic: IL-17A inhibitor
  Form: Solution for injection
  Route of administration: Subcutaneous (SC)
Drug: Placebo to izokibep — Form: Solution for injection
  Route of administration: Subcutaneous (SC)
  Arms: Group 1; Group 3; Group 4

SUMMARY:
Izokibep is a potent and selective inhibitor of interleukin (IL)-17A that is being developed for treatment of psoriatic arthritis (PsA).

This study will evaluate the efficacy of izokibep in subjects with PsA.

ELIGIBILITY:
Inclusion Criteria:

General

* Subject has provided signed informed consent including consenting to comply with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Subject must be ≥18 (or the legal age of consent in the jurisdiction in which the study is taking place) and ≤75 years of age, at the time of signing the informed consent.

Type of Subject and Disease Characteristics

* Clinical diagnosis of psoriatic arthritis (PsA) with symptom onset at least 6 months prior to first dose of study drug and fulfillment of the ClASsification for Psoriatic ARthritis (CASPAR) criteria at Screening.
* Active PsA defined as ≥3 tender joints (based on 68 joint counts) and ≥3 swollen joints (based on 66 joint counts) at Screening and Baseline Visits
* Rheumatoid factor (RF) and anti-cyclic citrullinated peptide (anti-CCP) negative at screening.
* Subject must have had an inadequate response, intolerance, or contraindication to at least one of the following:

  1. nonsteroidal anti-inflammatory drug (NSAID)
  2. conventional-synthetic disease-modifying anti-rheumatic drugs (csDMARD) (i.e. methotrexate, sulfasalazine, leflunomide, hydroxychloroquine, cyclosporine A)
  3. tumor necrosis factor-alpha inhibitor(s) (TNFi) (e.g. adalimumab, infliximab, etanercept, golimumab, certolizumab).
* For subjects using methotrexate, leflunomide, sulfasalazine, hydroxychloroquine, or apremilast, treated for ≥3 months and a stable dose (not to exceed 25 mg methotrexate per week, 20 mg leflunomide per day, sulfasalazine 3 g per day, hydroxychloroquine 400 mg per day, or apremilast 60 mg per day) for ≥4 weeks prior to first dose of study drug.
* For subjects using corticosteroids, must have been on a stable dose and regimen and not to exceed 7.5 mg per day of prednisone (or other corticosteroid equivalent to 7.5 mg per day of prednisone) for ≥4 weeks prior to first dose of study drug.
* Subjects using NSAIDs, or low potency opioid medications (tramadol, paracetamol in combination with hydrocodone or with codeine) must have been on a stable dose and regimen for ≥2 weeks prior to first dose of study drug.

Other Inclusions

* No known history of active tuberculosis (TB).
* Subject has a negative TB test at screening

Exclusion Criteria:

Disease-related Medical Conditions

* Any history or current confirmed diagnosis of inflammatory bowel disease (IBD)

OR

* Any of the following symptoms (of unknown etiology) or any signs or symptoms within the last year that in the opinion of the Investigator may be suggestive of IBD, with fecal calprotectin ≥ 500 μg/g; OR if fecal calprotectin >150 to <500 μg/g without confirmed approval from a GI consult that an IBD diagnosis is clinically unlikely when the following clinical signs and symptoms are present:

  1. prolonged or recurrent diarrhea
  2. prolonged or recurrent abdominal pain
  3. blood in stool
* History of fibromyalgia, or any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than psoriatic arthritis (PsA) (including, but not limited to rheumatoid arthritis, gout, connective tissue diseases). Prior history of axial spondyloarthritis or fibromyalgia is permitted if documentation of change in diagnosis to PsA or documentation that the diagnosis was made incorrectly. Prior history of reactive arthritis or axial spondyloarthritis is permitted if an additional diagnosis of PsA is made. Chronic osteoarthritis symptoms that in the Investigator's opinion may interfere with study assessments.
* Uncontrolled, clinically significant system disease
* Malignancy within 5 years
* Severe, uncontrolled, medically unstable mood disorder, such as severe depression.
* History or evidence of any clinically significant disorder (including psychiatric), condition, or disease that, in the opinion of the investigator, may pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Active infection or history of certain infections
* Candida infection requiring systemic treatment within 3 months prior to first dose of study drug.
* Tuberculosis or fungal infection seen on available chest x-ray taken within 3 months prior to first dose of study drug or at screening (Exception: documented evidence of completed treatment and clinically resolved).
* Known history of human immunodeficiency virus (HIV) or positive HIV test at screening.

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shepard Mpofu, MD, Clinical Development, Study Director — ACELYRIN Inc.
Locations (68):
- United States (40):
  - Clinical Research Site, Flagstaff, Arizona
  - Clinical Research Site, Glendale, Arizona
  - Clinical Research Site, Mesa, Arizona
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Tucson, Arizona
  - Clinical Research Site, Jonesboro, Arkansas
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Fountain Valley, California
  - Clinical Research Site, Fullerton, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Rancho Mirage, California
  - Clinical Research Site, Sacramento, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Santa Monica, California
  - Clinical Research Site, Upland, California
  - Clinical Research Site, Aventura, Florida
  - Clinical Research Site, Clearwater, Florida
  - Clinical Research Site, Kissimmee, Florida
  - Clinical Research Site, New Port Richey, Florida
  - Clinical Research Site, Ormond Beach, Florida
  - Clinical Research Site, Sarasota, Florida
  - Clinical Research Site, Gainesville, Georgia
  - Clinical Research Site, Hinsdale, Illinois
  - Clinical Research Site, Orland Park, Illinois
  - Clinical Research Site, Skokie, Illinois
  - Clinical Research Site, Lexington, Kentucky
  - Clinical Research Site, Grand Blanc, Michigan
  - Clinical Research Site, Kalispell, Montana
  - Clinical Research Site, Santa Fe, New Mexico
  - Clinical Research Site, Hickory, North Carolina
  - Clinical Research Site, Middleburg Heights, Ohio
  - Clinical Research Site, Corvallis, Oregon
  - Clinical Research Site, Duncansville, Pennsylvania
  - Clinical Research Site, Jackson, Tennessee
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Colleyville, Texas
  - Clinical Research Site, Irving, Texas
  - Clinical Research Site, Mesquite, Texas
  - Clinical Research Site, Seattle, Washington
  - Clinical Research Site, Beckley, West Virginia
- Bulgaria (4):
  - Clinical Research Site, Burgas
  - Clinical Research Site, Pleven
  - Clinical Research Site, Rousse
  - Clinical Research Site, Sofia
- Canada (5):
  - Clinical Research Site, Sydney, Nova Scotia
  - Clinical Research Site, Windsor, Ontario
  - Clinical Research Site, Québec, Quebec
  - Clinical Research Site, Trois-Rivières, Quebec
  - Clinical Research Site, Saskatoon, Saskatchewan
- Czechia (3):
  - Clinical Research Site, Ostrava
  - Clinical Research Site, Prague
  - Clinical Research Site, Zlín
- Germany (2):
  - Clinical Research Site, Frankfurt am Main
  - Clinical Research Site, Hamburg
- Hungary (5):
  - Clinical Research Site, Budapest
  - Clinical Research Site (003), Budapest
  - Clinical Research Site, Kalocsa
  - Clinical Research Site, Székesfehérvár
  - Clinical Research Site, Veszprém
- Poland (6):
  - Clinical Research Site, Bialystok
  - Clinical Research Site, Bydgoszcz
  - Clinical Research Site, Elblag
  - Clinical Research Site, Krakow
  - Clinical Research Site, Poznan
  - Clinical Research Site, Warsaw
- Spain (3):
  - Clinical Research Site, Alcobendas
  - Clinical Research Site, Santiago de Compostela
  - Clinical Research Site, Seville

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 351 participants with Psoriatic Arthritis (PsA) symptoms were recruited in Canada, United States, Bulgaria, Czech Republic, Germany, Hungary, Poland, and Spain between November 2022 and August 2024.
Pre-assignment Details: This study was divided into two Periods. In Period 1 (Phase 2b portion of the study), participants received either izokibep or placebo, until Week 16. Period 2 (Phase 3 portion of the study) lasted until Week 52. Participants who received placebo QW during Period 1 started receiving izokibep QW during Period 2 and participants who received izokibep during Period 1 continued to receive izokibep at the same dosing frequency in Period 2.
Groups:
- Period 1: Placebo QW ; Period 2: Izokibep 160 mg QW: Participants received placebo as a subcutaneous (SC) injection QW for up to Week 16. Then, participants received izokibep 160 mg as a SC injection QW from Week 16 up to Week 52.
- Izokibep 80 mg Q4W: Participants received izokibep 80 mg as a SC injection every 4 weeks (Q4W) for up to Week 52. Matching placebo QW was administered for weeks in-between izokibep to maintain the blind.
- Izokibep 160 mg Q2W: Participants received izokibep 160 mg as a SC injection every Q2W for up to Week 52. Matching placebo QW was administered for weeks in-between izokibep to maintain the blind.
- Izokibep 160 mg QW: Participants received izokibep 160 mg as a SC injection QW for up to Week 52.
Period: Overall Study
Arm/Group | Period 1: Placebo QW ; Period 2: Izokibep 160 mg QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Started | 118 | 8 | 113 | 112
Completed Period 1 | 114 | 8 | 111 | 105
Completed | 64 | 4 | 57 | 52
Not Completed | 54 | 4 | 56 | 60
Not completed — Withdrawal by Subject | 14 | 0 | 9 | 20
Not completed — Lost to Follow-up | 3 | 0 | 7 | 2
Not completed — Termination of Study By Sponsor | 37 | 4 | 40 | 38

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all participants randomized who received at least one administration of test material was included in the summaries and analyses.
Groups:
- Period 1: Placebo QW: Participants received placebo as a SC injection QW up to Week 16.
- Izokibep 80 mg Q4W: Participants received izokibep 80 mg as a SC injection every 4 weeks (Q4W) up to Week 52. Matching placebo QW was administered for weeks in-between izokibep to maintain the blind.
- Izokibep 160 mg Q2W: Participants received izokibep 160 mg as a SC injection every Q2W up to Week 52. Matching placebo QW was administered for weeks in-between izokibep to maintain the blind.
- Izokibep 160 mg QW: Participants received izokibep 160 mg as a SC injection QW up to Week 52.
- Total: Total of all reporting groups
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW | Total
Number analyzed (Participants) | 118 | 8 | 113 | 112 | 351
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (11.74) | 63.1 (9.40) | 49.5 (13.26) | 51.8 (12.20) | 51.6 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 5 | 46 | 48 | 166
  Male | 51 | 3 | 67 | 64 | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 1 | 14 | 7 | 35
  Not Hispanic or Latino | 105 | 7 | 99 | 104 | 315
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 2 | 7
  White | 110 | 8 | 108 | 109 | 335
  More than one race | 0 | 0 | 0 | 0 | 0
  Other | 2 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved 50% Improvement in American College of Rheumatology (ACR50) at Week 16
Description: ACR50 is a clinical trial measure for PsA, indicating a 50% improvement in symptoms. To qualify, participants must show a 50% reduction in tender and swollen joint counts plus improvements in three of five additional criteria, including pain, global assessments, physical function, and inflammatory markers. ACR50 is binary-patients either meet it or not.
Time Frame: Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: Placebo QW: Participants received placebo as SC injection QW for up to Week 16.
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 118 | 8 | 113 | 112
Participants | 18 | 4 | 49 | 45
Statistical Analysis 1: Comparison: Period 1: Placebo QW vs Izokibep 80 mg Q4W; Test type: Superiority; p = 0.0377, Cochran-Mantel-Haenszel; Risk Difference (RD) = 36.22, Standard Error of Mean 17.43
Statistical Analysis 2: Comparison: Period 1: Placebo QW vs Izokibep 160 mg Q2W; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 27.69, Standard Error of Mean 5.68
Statistical Analysis 3: Comparison: Period 1: Placebo QW vs Izokibep 160 mg QW; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.44, Standard Error of Mean 5.65

2. Secondary Outcome: Number of Participants With Baseline ≥ 3% Body Surface Area (BSA) Psoriasis Who Achieved a 90% or Greater Reduction in Psoriasis Area and Severity Index (PASI90) at Week 16
Description: PASI is a tool used in clinical trials to measure the severity and extent of psoriasis. Scores range from a minimum of 0 to a maximum of 72, with higher scores indicating more severe disease.
Time Frame: Baseline and Week 16
Population: Full Analysis Set: all participants randomized who received at least one administration of test material was included in the summaries and analyses.
  Only participants with ≥ 3% BSA psoriasis at baseline were analyzed for this endpoint.
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: Placebo QW: Participants received placebo as a SC injection QW for up to Week 16.
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 60 | 5 | 64 | 59
Participants | 7 | 3 | 37 | 38
Statistical Analysis 1: Comparison: Period 1: Placebo QW vs Izokibep 80 mg Q4W; Test type: Superiority; p = 0.0483, Cochran-Mantel-Haenszel; Risk Difference (RD) = 43.71, Standard Error of Mean 22.14
Statistical Analysis 2: Comparison: Period 1: Placebo QW vs Izokibep 160 mg Q2W; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 46.15, Standard Error of Mean 7.62
Statistical Analysis 3: Comparison: Period 1: Placebo QW vs Izokibep 160 mg QW; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 52.80, Standard Error of Mean 7.56

3. Secondary Outcome: Number of Participants With Baseline Enthesitis > 0 With Resolution of Enthesitis (Leeds Enthesitis Index [LEI] = 0) at Week 16
Description: LEI is a clinical tool used to assess enthesitis in conditions like psoriatic arthritis and spondyloarthritis. It evaluates six sites: bilateral lateral epicondyles, medial femoral condyles, and achilles tendons. Each site is scored 0 (no pain) or 1 (pain on pressure), with a total score ranging from a minimum of 0 to a maximum of 6, where higher scores indicate more severe enthesitis.
Time Frame: Baseline and Week 16
Population: Full Analysis Set: all participants randomized who received at least one administration of test material was included in the summaries and analyses.
  Only participants with LEI > 0 at baseline were analyzed for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 75 | 5 | 68 | 66
Participants | 35 | 4 | 38 | 30
Statistical Analysis 1: Comparison: Period 1: Placebo QW vs Izokibep 80 mg Q4W; Test type: Superiority; p = 0.0883, Cochran-Mantel-Haenszel; Risk Difference (RD) = 32.26, Standard Error of Mean 18.93
Statistical Analysis 2: Comparison: Period 1: Placebo QW vs Izokibep 160 mg Q2W; Test type: Superiority; p = 0.2713, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.19, Standard Error of Mean 8.35
Statistical Analysis 3: Comparison: Period 1: Placebo QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.8872, Cochran-Mantel-Haenszel; Risk Difference (RD) = -1.20, Standard Error of Mean 8.44

4. Secondary Outcome: Number of Participants Achieving Minimal Disease Activity (MDA) at Week 16
Description: A participants was classified as being in MDA when at least five of the following seven criteria were met:
  * Tender joint count based on 68 joints (TJC68) ≤ 1
  * Swollen joint count based on 66 joints (SJC66) ≤ 1
  * PASI ≤ 1 or BSA ≤ 3%
  * Participant's Pain Assessment (Visual Analogue Scale [VAS]) ≤ 15 mm
  * Participant's Global Activity VAS ≤ 20 mm (corresponding to participant's Global Assessment of Disease Activity)
  * Health Assessment Questionnaire-Disability Index (HAQ-DI) ≤ 0.5
  * Tender enthesitis points ≤ 1 out of 6 sites assessed by the LEI.
Time Frame: Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 118 | 8 | 113 | 112
Participants | 17 | 3 | 47 | 46
Statistical Analysis 1: Comparison: Period 1: Placebo QW vs Izokibep 80 mg Q4W; Test type: Superiority; p = 0.1654, Cochran-Mantel-Haenszel; Risk Difference (RD) = 23.45, Standard Error of Mean 16.90
Statistical Analysis 2: Comparison: Period 1: Placebo QW vs Izokibep 160 mg Q2W; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.58, Standard Error of Mean 5.53
Statistical Analysis 3: Comparison: Period 1: Placebo QW vs Izokibep 160 mg QW; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.84, Standard Error of Mean 5.55

5. Secondary Outcome: Number of Participants Achieving 20% Improvement in ACR (ACR20) at Week 16
Description: ACR20 is a clinical trial measure for PsA, indicating a 20% improvement in symptoms. To qualify, participants must show a 20% reduction in tender and swollen joint counts plus improvements in three of five additional criteria, including pain, global assessments, physical function, and inflammatory markers. ACR20 is binary-patients either meet it or not.
Time Frame: Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: Placebo QW: Participants received placebo as a SC injection QW for up to 16 Week.
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 118 | 8 | 113 | 112
Participants | 41 | 6 | 72 | 66
Statistical Analysis 1: Comparison: Period 1: Placebo QW vs Izokibep 80 mg Q4W; Test type: Superiority; p = 0.0106, Cochran-Mantel-Haenszel; Risk Difference (RD) = 43.09, Standard Error of Mean 16.85
Statistical Analysis 2: Comparison: Period 1: Placebo QW vs Izokibep 160 mg Q2W; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.46, Standard Error of Mean 6.22
Statistical Analysis 3: Comparison: Period 1: Placebo QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Risk Difference (RD) = 23.70, Standard Error of Mean 6.40

6. Secondary Outcome: Number of Participants With Baseline Psoriatic Arthritis Impact of Disease (PsAID) Score ≥ 3 With Improvement in PsAID Score at Week 16
Description: The PsAID consists of nine items, each scored on a numeric rating scale (0-10), covering key aspects of disease burden, including pain, fatigue, skin problems, work/leisure activities, functional capacity, sleep disturbance, anxiety, coping, and social participation. The total score is calculated as a weighted sum of these individual items, with higher scores indicating a greater impact of the disease. The minimum score is 0 (no disease impact), while the maximum is 10 (worst possible disease impact). Reaching an improvement was considered an increase of 3 units from baseline score.
Time Frame: Week 16
Population: Full Analysis Set: all participants randomized who received at least one administration of test material was included in the summaries and analyses.
  Only participants with PsAID ≥ 3 at baseline were analyzed for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 98 | 7 | 102 | 105
Participants | 12 | 3 | 43 | 40
Statistical Analysis 1: Comparison: Period 1: Placebo QW vs Izokibep 80 mg Q4W; Test type: Superiority; p = 0.1147, Cochran-Mantel-Haenszel; Risk Difference (RD) = 30.15, Standard Error of Mean 19.11
Statistical Analysis 2: Comparison: Period 1: Placebo QW vs Izokibep 160 mg Q2W; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.04, Standard Error of Mean 5.92
Statistical Analysis 3: Comparison: Period 1: Placebo QW vs Izokibep 160 mg QW; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.99, Standard Error of Mean 5.81

7. Secondary Outcome: Change in Physical Function as Assessed by HAQ-DI From Baseline to Week 16
Description: The HAQ-DI consists of 20 questions divided into eight categories: dressing, arising, eating, walking, hygiene, reaching, grip, and other activities. Each item is scored on a scale from 0 to 3, where 0 = no difficulty, 1 = some difficulty, 2 = much difficulty, and 3 = unable to perform. The final HAQ-DI score is calculated as the average of the highest scores in each category, resulting in a range from 0 (no disability) to 3 (severe disability). Higher scores indicate greater functional impairment. A negative change indicates an improvement in functional impairment.
Time Frame: Baseline and Week 16
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 114 | 8 | 106 | 103
Score on scale | -0.14 [-0.23 to -0.06] | -0.03 [-0.35 to 0.28] | -0.30 [-0.39 to -0.21] | -0.31 [-0.40 to -0.22]
Statistical Analysis 1: Comparison: Period 1: Placebo QW vs Izokibep 80 mg Q4W; Test type: Superiority; p = 0.514, Mixed model repeated measures analysis; LS Mean Difference = 0.11, 95% CI 2-sided [-0.22 to 0.44], Standard Error of Mean 0.166
Statistical Analysis 2: Comparison: Period 1: Placebo QW vs Izokibep 160 mg Q2W; Test type: Superiority; p = 0.010, Mixed model repeated measures analysis; LS Mean Difference = -0.16, 95% CI 2-sided [-0.28 to -0.04], Standard Error of Mean 0.061
Statistical Analysis 3: Comparison: Period 1: Placebo QW vs Izokibep 160 mg QW; Test type: Superiority; p = 0.006, Mixed model repeated measures analysis; LS Mean Difference = -0.17, 95% CI 2-sided [-0.29 to -0.05], Standard Error of Mean 0.061

8. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and AE of Special Interest During Period 1
Description: An AE was any untoward medical occurrence in a participant, regardless of a causal relationship with the study treatment. TEAEs included any event occurring after the participant received study treatment. Clinically significant changes in vital signs, electrocardiograms and laboratory tests recorded after treatment administration were documented as TEAEs.
  TEAEs were considered serious if they led to death, were life-threatening, required hospitalization or its prolongation, caused disability, resulted in congenital anomalies or were considered medically important.
  The events of special interest monitored were : candida infection; inflammatory bowel disease; suicidal ideation; malignancies; major adverse cardiovascular and cerebrovascular events (cerebrovascular accident and transient ischemic attack, nonfatal myocardial infarction or unstable angina, cardiovascular death); tuberculosis; infections (opportunistic, serious, or fungal); cytopenia; systemic hypersensitivity reactions.
Time Frame: Up to Week 16, or 4 weeks after participant's last dose in case of treatment discontinuation
Population: Safety Analysis Set: All participants randomized who received at least one administration of test material during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Placebo QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 118 | 8 | 113 | 112
Participants
  TEAEs | 48 | 6 | 76 | 82
  Serious TEAEs | 1 | 2 | 2 | 3
  AEs of Special Interest | 2 | 1 | 5 | 6

9. Secondary Outcome: Number of Participants Who Experienced TEAEs, Serious TEAEs and AE of Special Interest During Period 2
Description: as for outcome 8
Time Frame: First dose of study treatment on or after Week 16 up to Week 55
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Period 2: Placebo/Izokibep 160 mg QW: Participants received izokibep 160 mg as a SC injection QW from Week 16 up to Week 52.
Arm/Group | Period 2: Placebo/Izokibep 160 mg QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 114 | 8 | 103 | 98
Participants
  TEAEs | 89 | 5 | 67 | 67
  Serious TEAEs | 4 | 1 | 7 | 2
  AEs of Special Interest | 3 | 1 | 5 | 2

10. Secondary Outcome: Number of Participants With a Positive Treatment-emergent Anti-drug Antibody (ADA) Result
Description: Blood samples were collected at different timepoints throughout the study. ADA is considered "Positive" if any titer value is available.
Time Frame: Baseline to Week 65
Population: ADA Analysis Set: Included all participants include who received at least one administration of izokibep and had both a baseline ADA measurement and at least one post-dose ADA measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Period 1: Placebo QW; Period 2: Izokibep 160 mg QW: Participants received placebo as a SC injection QW for up to Week 16. Then, participants received izokibep 160 mg as a SC injection QW from Week 16 up to Week 52.
Arm/Group | Period 1: Placebo QW; Period 2: Izokibep 160 mg QW | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
Number analyzed (Participants) | 116 | 8 | 108 | 108
Participants
  Baseline | 56 | 4 | 57 | 54
  Week 2: number analyzed (Participants) | 113 | 8 | 105 | 105
  Week 2 | 56 | 3 | 61 | 54
  Week 4: number analyzed (Participants) | 114 | 8 | 105 | 106
  Week 4 | 56 | 4 | 58 | 55
  Week 12: number analyzed (Participants) | 114 | 6 | 106 | 103
  Week 12 | 53 | 2 | 55 | 51
  Week 16: number analyzed (Participants) | 112 | 8 | 103 | 100
  Week 16 | 54 | 6 | 57 | 57
  Week 24: number analyzed (Participants) | 104 | 8 | 102 | 96
  Week 24 | 40 | 5 | 70 | 75
  Week 36: number analyzed (Participants) | 102 | 8 | 97 | 93
  Week 36 | 62 | 7 | 67 | 76
  Week 52: number analyzed (Participants) | 83 | 7 | 87 | 76
  Week 52 | 65 | 7 | 63 | 68
  Follow-up Visit - Week 59: number analyzed (Participants) | 96 | 8 | 92 | 87
  Follow-up Visit - Week 59 | 76 | 6 | 67 | 77
  End of Study - Week 65: number analyzed (Participants) | 64 | 3 | 52 | 49
  End of Study - Week 65 | 49 | 2 | 31 | 40

ADVERSE EVENTS:
Time Frame: For Placebo QW - Period 1: Up to Week 16, or 4 weeks after participant's last dose in case of treatment discontinuation. A TEAE that occurred before the first dose of study drug in Period 2 and is within 28 days after the end of study drug in Period 1 is assigned to Period 1. For Placebo/Izokibep 160 mg QW - Period 2: From Week 16 up to Week 55. For Izokibep 80 mg Q4W, Izokibep 160 mg Q2W, Izokibep 160 mg QW: Up to Week 55.
Description: Safety Analysis Set: All participants randomized who received at least one administration of test material during the study.
Groups:
- Placebo QW - Period 1: Participants received placebo as a SC injection QW for up to Week 16.
- Placebo/Izokibep 160 mg QW - Period 2: Participants received izokibep 160 mg as a SC injection QW from Week 16 up to Week 52.
Arm/Group | Placebo QW - Period 1 | Placebo/Izokibep 160 mg QW - Period 2 | Izokibep 80 mg Q4W | Izokibep 160 mg Q2W | Izokibep 160 mg QW
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/114 | 0/8 | 0/113 | 0/112
Serious Adverse Events (participants affected / at risk) | 1/118 | 4/114 | 2/8 | 8/113 | 4/112
Other Adverse Events (participants affected / at risk) | 9/118 | 65/114 | 6/8 | 78/113 | 84/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QW - Period 1 (N=118) | Placebo/Izokibep 160 mg QW - Period 2 (N=114) | Izokibep 80 mg Q4W (N=8) | Izokibep 160 mg Q2W (N=113) | Izokibep 160 mg QW (N=112)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Periumbilical abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Wernicke-Korsakoff syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QW - Period 1 (N=118) | Placebo/Izokibep 160 mg QW - Period 2 (N=114) | Izokibep 80 mg Q4W (N=8) | Izokibep 160 mg Q2W (N=113) | Izokibep 160 mg QW (N=112)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 7 | 1 | 4 | 3
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 53 | 2 | 52 | 65
Injection site pruritus (General disorders) | 1 | 27 | 2 | 25 | 29
Injection site swelling (General disorders) | 0 | 13 | 1 | 13 | 13
Injection site pain (General disorders) | 1 | 8 | 0 | 8 | 8
Injection site rash (General disorders) | 0 | 0 | 1 | 8 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 7 | 2
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 14 | 0 | 18 | 13
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 2 | 10 | 20
COVID-19 (Infections and infestations) | 2 | 0 | 1 | 8 | 4
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 2 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT05623345/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT05623345/SAP_001.pdf